CLINICAL TRIAL: NCT03780556
Title: Lornoxicam With Low Dose Ketamine Versus Pethidine to Control Pain of Acute Renal Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASU 5418
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Renal Colic
Keywords: Renal pain; lornoxicam; pethidine; emergency room; ketamine
MeSH Terms: conditions — Renal Colic; Emergencies | interventions — lornoxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lornixicam (Active Comparator): Patients received lornoxicam 8 mg intravenous to control pain
  Interventions: Drug: Lornoxicam and mepridine
- Pethidine (Active Comparator): Patients received pethidine 50mg intravenous to control pain
  Interventions: Drug: Lornoxicam and mepridine

INTERVENTIONS:
Drug: Lornoxicam and mepridine — compare the effect of each to control pain

SUMMARY:
Patients with acute renal colic divided into 2 groups. Group L administered ornoxicam and Group P administered pethidine and VAS was recorded for both groups.

DETAILED DESCRIPTION:
Prospective, randomized, double blind clinical study including 120 patients with acute renal pain admitted in emergency department. They were randomly assigned to one of two groups using a computer-generated table. Group L received lornoxicam 8 mg IV plus 0.15 mg.kg-1 ketamine and Group P received pethidine 50 mg IV. Parameters were observed at baseline and after 0, 15, 30, 45 and 1 hour of drug treatment. The efficacy of the drug was measured by observing: patient rated pain, time to pain relief, rate of pain recurrence, the need for rescue analgesia, adverse events and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who did not administer any analgesics at least within the last two hours. - -
* Patients aged between 20-60 years.

Exclusion Criteria:

* Patients with previous renal surgery
* liver and renal failure
* hypersensitivity to lornoxicam, ketamine and pethidine, history of peptic ulcer,
* gastrointestinal bleeding and perforation,
* hypertensive and history of cardiac diseases
* pregnancy and lactation and
* urine examination showing more than 5 leukocytes suggestive of pyuria.
* patients with hyperthyroidism are excluded

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in pain feeling | 0hours, 1hour,2hours,3hours,4hours after drug administration in both groups
  We assess this through Visual analogue scale score to assess pain due to renal colic, number 10 means maximum pain feeling and 0 means no pain at all.
No need for more analgesics | Registration of analgesic needed for 12h after the attack
  Rescue analgesics administration

CONTACTS AND LOCATIONS:
Locations (1):
- ِAin Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No